CLINICAL TRIAL: NCT06946914
Title: Misoprostol Administration Before Elective Caesarean Section to Reduce the Risk of Respiratory Morbidity in Newborns
Brief Title: Misoprostol Before Caesarean Section
Acronym: Miso/CS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Merna Ashraf Ahmed Farid, gynaecologist and obsteterician resident, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KFSIRB200-244
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Misoprostol; Respiratory Distress Syndrome (RDS) of Neonate; Caesarean Section
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Misoprostol before elective cesarean section . (Active Comparator): candidates will receive 100mcg Misoprostol one hour before elective caesarean section.
  Interventions: Drug: Misoprostol
- Giving no treatment before elective caesarean section. (Placebo Comparator): candidates will receive no treatment before elective caesarean section.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — administration of 100mg of misoprostol to evaluate the efficacy of Misoprostol before elective cesarean section in pregnant women with gestational age less than 38 weeks for preventing the occurrence of neonatal respiratory morbidity.

SUMMARY:
The aim of our study is to evaluate the efficacy of Misoprostol before elective cesarean section in pregnant women with gestational age less than 38 weeks for preventing the occurrence of neonatal respiratory morbidity.

DETAILED DESCRIPTION:
Caesarean section is one of the most common carried out surgical procedures in modern obstetrics. About 18.5 million caesarean section are conducted yearly worldwide, and 21-33% of all caesarean section are performed in middle and high-income countries.

The most frequent complications that are seen in neonates include respiratory morbidity, hypoglycemia, sepsis, and admission to the neonatal intensive care unit (NICU). The family and caregivers are affected in many ways when a newborn is admitted to the intensive care unit.

Both preterm and term infants delivered by caesarean section have been reported to experience respiratory distress syndrome, which is brought on by a surfactant deficiency.

Respiratory distress (RD) affects about 27% of babies born, and it is more common in newborns delivered by elective cesarean section (ECS) than in emergency CS or vaginally.

In the neonatal intensive care unit, neonatal respiratory distress syndrome (NRDS), which is mostly brought on by pulmonary surfactant insufficiency after delivery, is acknowledged as one of the most frequent causes of respiratory distress in newborn preterm infants.

In babies with NRDS, pulmonary insufficiency begins after birth and gets worse throughout the course of the first two days of life. Pulmonary surfactant, secreted by type 2 pneumocytes at about 24 weeks gestation, reaches a level that facilitates breathing after birth at 36 weeks.

Misoprostol, an oral medication, an analogue of PGE1, was created and introduced to treat and prevent upper gastrointestinal ulcers caused by nonsteroidal anti-inflammatory drugs (NSAIDs). Use during pregnancy was not advised because of its uterotonic impact.

Misoprostol was originally licensed for oral use; however, vaginal and sublingual routes of administration are becoming more and more popular supported by pharmacokinetic studies focusing on the systemic bioavailability parameters achieved. While the sublingual route seems to have the greater bioavailability and safety.

Misoprostol's characteristics include being cheap and easily stored at room temperature (shelf life: 3 years). It can be used safely in individuals with hypertension and asthma because, as compared to other prostaglandins, it has less impact on the smooth muscle of the bronchi and cardiovascular system. It is not impacted by the outside temperature and doesn't require syringes, needles, or refrigeration for administration or storage, respectively.

Misoprostol is known as a safe drug with very few side effects. Menstrual cramps, fever, chills, shivering, diarrhea, headaches, and abdominal pain are among its frequent side effects.

Prostaglandins are substances that have been successfully used for labor induction in the pregnant females and the E series being preferred over others due to the fact that they are more utero selective. It was found that prostaglandin has beneficial effects on the neonatal lungs as it causes the reabsorption of lung fluid from the fetal lung and promotes surfactant secretion by inducing the catecholamine surge. However on clinical practice, the effectiveness of the antenatal prophylactic administration prostaglandin on reducing the neonatal respiratory morbidity is still not clear.

Prior studies reported an option for reducing surgical bleeding and their results showed agreement that oxytocin prevented postpartum hemorrhage by helping the uterine contraction. Furthermore, administration of other uterotonic agents have been studied for more effectiveness of treating excessive blood loss. Misoprostol, a prostaglandin E1 analogue, shows a good uterotonic property and less side effects which is available in worldwide even in the low resource setting.

Systematic reviews also demonstrated that misoprostol combined with oxytocin decreased the incidence of PPH significantly. According to their synergistic effects which oxytocin acts immediately with short half-life while misoprostol provides sustainable efficacy of uterine contractility. Misoprostol, in a tablet preparation, can be prescribed in different route including sublingual, oral, rectal and vaginal. In addition, intrauterine insertion is well documented in many studies recently. While an optimal dosage of intrauterine route has not been well established, range of dosage from 400 to 800 μg were used safely. However, side effect such as pyrexia (body temperature ≥ 38 ◦C) was significant high related to higher doses (≥800 μg) of misoprostol was reported .

Various studies have been carried out regarding the incidence and associated factors of respiratory distress in preterm neonates. Such research will be crucial in helping to enhance treatment protocols and raise the infant survival rate, particularly for those neonates who are most at risk of dying from preterm complications like respiratory distress.

ELIGIBILITY:
Inclusion Criteria:

* Women with indication for elective caesarean section.
* Age less than 35 years old.
* Gestational age less than 38 weeks.
* Gestational age will be confirmed by certain LMP or reliable early ultrasound measurement of crown-rump length.
* Singleton pregnancy with no major anomalies

Exclusion Criteria:

* Any obstetric disorders as preeclampsia and diabetes.
* Fetus with oligohydramnios, intrauterine growth restriction.
* Any contraindications to misoprostol like those with previous allergic reaction or hypersensitivity to prostaglandin hemorrhagic disorders, and severe anemia.
* History of more than or equal 2 previous caesarean section.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of Transient tachypnea of the newborn which defined by increase respiratory rate more than 60 cycle per minute in pregnant women with gestational age less than 38 weeks before elective cesarean section | in the first 5 minute after delivery of fetus post operative

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr El-sheikh University Hospital, Kafr Ash Shaykh, Egypt, Egypt